CLINICAL TRIAL: NCT05961722
Title: The Effect of Choosing of Preoperative Intravenous Fluid Type on the Postoperative Nausea, Vomiting, Anxiety and Pain After Laparoscopic Cholecystectomy
Brief Title: Preoperative Intravenous Fluid Type and Postoperative Nausea
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AnkaraEtlikYusufOzguner003
Record Dates: First submitted 2023-07-13; First posted 2023-07-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post Operative Pain; Nausea and Vomiting, Postoperative; Anxiety
Keywords: preoperative intravenous fluid type; laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Anxiety Disorders | interventions — Sodium Chloride

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group receiving preoperative and intraoperative saline infusion.
  Interventions: Other: preoperative IV 0.9% saline 400 ml
- Group 2: The group receiving preoperative dextrose and intraoperative saline infusion.
  Interventions: Other: preoperative dextrose 5% 400 ml
- Group 3: The group receiving preoperative and intraoperative dextrose infusion.
  Interventions: Other: preoperative and intraoperative dextrose 5% 400 ml

INTERVENTIONS:
Other: preoperative IV 0.9% saline 400 ml — Group 1 will be infused with IV 0.9% saline 400 mL.
  Groups: Group 1
Other: preoperative dextrose 5% 400 ml — Group 2 will be infused with dextrose 5% Dekstroz 400 ml.
  Groups: Group 2
Other: preoperative and intraoperative dextrose 5% 400 ml — Group 3 will be infused with dextrose preoperative 200 ml and intraoperative 200 ml 5% dextrose infusion.
  Groups: Group 3

SUMMARY:
In this study, it was aimed to investigate the relationship between postoperative nausea and vomiting, anxiety levels and pain scores in the postoperative period according to dosing and choosing of intravenous fluid type that the patients received in the preoperative period.

DETAILED DESCRIPTION:
Fluid management is an integral and important part of perioperative treatment. In order to prevent organ damage, a key components of assuring adequate organ perfusion is to provide adequate volume and appropriate fluid. Types of the fluids, amount of the fluid given and timing of the administration are the main topics that determine the fluid management strategy. Colloids (e.g. albumin or fresh frozen plasma (FFP)) and crystalloids (e.g. ringer lactate, isotonic, 5% dextrose) are types of intravenous fluids that are used for fluid replacement apart from blood transfusion . Crystalloids are low-cost salt solutions with small molecules, which can move around easily when injected into the body.

There are studies reporting that fluid therapy applied in the preoperative period reduces gastric acid secretion and reduces stomach movements and nausea and vomiting. In addition, there are studies reporting that fluids given in the preoperative period have a positive effect on anxiety levels by reducing the feeling of hunger and thirst in patients. There are studies reporting that fluid therapy reduces ATP destruction and oxidative stress, which contributes to the reduction of pain levels.

90 ASA I-II patients who will undergo laparoscopic cholecystectomy surgery will be included in the study and will be divided into three equal groups. Patients in Group 1 were administered 400 ml 0.9% saline infusion within 30 minutes, 2 hours before surgery. Patients in Group 2 were infused with 400 ml 5% Dextrose at the same infusion rate. In groups 1 and 2, 10 ml/kg/h 0.9% saline infusion was applied during the intraoperative period. Patients in Group 3 were administered 200 ml dextrose infusion in the preoperative period and 200 ml dextrose infusion in the intraoperative period. 0.9% saline infusion was applied so that the total intraoperative fluid volume was the same as in the other groups.

Postoperative nausea and vomiting (PONV) , within 24 hours was compared between groups by PONV score. Other outcomes were the antiemetic drugs needed, The NRS Score, The State-Trait Anxiety Inventory , additional analgesic drug requirement.

In this study, it was aimed to investigate the relationship between postoperative nausea and vomiting, anxiety levels and pain scores in the postoperative period according to dosing and choosing of intravenous fluid type that the patients received in the preoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic cholecystectomy
* Patients over the age of 18

Exclusion Criteria:

* Patients who do not accept the study
* Diabetes Mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 90 ASA I-II patients who will undergo laparoscopic cholecystectomy surgery will be included in the study and will be divided into three equal groups.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
PONV Score | 0 hours postoperatively
  Postoperative nausea and vomitting recording in patients undergone laparoscopic cholocystectomy.
  * 0=no PONV: patient reports no nausea and has had no emesis episodes;
  * 1=mild PONV: patient reports nausea but declines antiemetic treatment;
  * 2=moderate PONV: patient reports nausea and accepts antiemetic treatment; and
  * 3=severe PONV: nausea with any emesis episode (retching or vomiting). Higher scores indicate severe postoperative nausea and vomitting.
PONV Score | 2 hours postoperatively
  Postoperative nausea and vomitting recording in patients undergone laparoscopic cholocystectomy.
  * 0=no PONV: patient reports no nausea and has had no emesis episodes;
  * 1=mild PONV: patient reports nausea but declines antiemetic treatment;
  * 2=moderate PONV: patient reports nausea and accepts antiemetic treatment; and
  * 3=severe PONV: nausea with any emesis episode (retching or vomiting). Higher scores indicate severe postoperative nausea and vomitting.
PONV Score | 4 hours postoperatively
  Postoperative nausea and vomitting recording in patients undergone laparoscopic cholocystectomy.
  * 0=no PONV: patient reports no nausea and has had no emesis episodes;
  * 1=mild PONV: patient reports nausea but declines antiemetic treatment;
  * 2=moderate PONV: patient reports nausea and accepts antiemetic treatment; and
  * 3=severe PONV: nausea with any emesis episode (retching or vomiting). Higher scores indicate severe postoperative nausea and vomitting.
PONV Score | 8 hours postoperatively
  Postoperative nausea and vomitting recording in patients undergone laparoscopic cholocystectomy.
  * 0=no PONV: patient reports no nausea and has had no emesis episodes;
  * 1=mild PONV: patient reports nausea but declines antiemetic treatment;
  * 2=moderate PONV: patient reports nausea and accepts antiemetic treatment; and
  * 3=severe PONV: nausea with any emesis episode (retching or vomiting). Higher scores indicate severe postoperative nausea and vomitting.
PONV Score | 12 hours postoperatively
  Postoperative nausea and vomitting recording in patients undergone laparoscopic cholocystectomy.
  * 0=no PONV: patient reports no nausea and has had no emesis episodes;
  * 1=mild PONV: patient reports nausea but declines antiemetic treatment;
  * 2=moderate PONV: patient reports nausea and accepts antiemetic treatment; and
  * 3=severe PONV: nausea with any emesis episode (retching or vomiting). Higher scores indicate severe postoperative nausea and vomitting.
PONV Score | 24 hours postoperatively
  Postoperative nausea and vomitting recording in patients undergone laparoscopic cholocystectomy.
  * 0=no PONV: patient reports no nausea and has had no emesis episodes;
  * 1=mild PONV: patient reports nausea but declines antiemetic treatment;
  * 2=moderate PONV: patient reports nausea and accepts antiemetic treatment; and
  * 3=severe PONV: nausea with any emesis episode (retching or vomiting). Higher scores indicate severe postoperative nausea and vomitting.

SECONDARY OUTCOMES:
Pain on the Numeric Rating Scale (NRS) | 0 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 2 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 4 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 8 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 12 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
Pain on the Numeric Rating Scale (NRS) | 24 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.
State-Trait Anxiety Inventory ( The STAI ) | 2 hours before induction of anesthesia
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
State-Trait Anxiety Inventory ( The STAI ) | 0 hours postoperatively
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoorn EJ. Intravenous fluids: balancing solutions. J Nephrol. 2017 Aug;30(4):485-492. doi: 10.1007/s40620-016-0363-9. Epub 2016 Nov 29. PMID 27900717
- [Result] Agarwal A, Dhiraaj S, Tandon M, Singh PK, Singh U, Pawar S. Evaluation of capsaicin ointment at the Korean hand acupressure point K-D2 for prevention of postoperative nausea and vomiting. Anaesthesia. 2005 Dec;60(12):1185-8. doi: 10.1111/j.1365-2044.2005.04402.x. PMID 16288616
- [Result] Hausel J, Nygren J, Lagerkranser M, Hellstrom PM, Hammarqvist F, Almstrom C, Lindh A, Thorell A, Ljungqvist O. A carbohydrate-rich drink reduces preoperative discomfort in elective surgery patients. Anesth Analg. 2001 Nov;93(5):1344-50. doi: 10.1097/00000539-200111000-00063. PMID 11682427
- [Result] Kristoffersen L, Malahleha M, Duze Z, Tegnander E, Kapongo N, Stoen R, Follestad T, Eik-Nes SH, Bergseng H. Randomised controlled trial showed that neonates received better pain relief from a higher dose of sucrose during venepuncture. Acta Paediatr. 2018 Dec;107(12):2071-2078. doi: 10.1111/apa.14567. Epub 2018 Oct 2. PMID 30188590